CLINICAL TRIAL: NCT00412659
Title: An Expertise-based Randomized Controlled Trial Comparing Midline Excision Versus Karydakis Operation at Surgery for Pilonidal Sinus
Brief Title: Mid-line Excision Versus Karydakis Operation for Pilonidal Sinus
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: County Council of Norrbotten, Sweden (Other Government); Norrlandstingens Regionförbund (Other)
Responsible Party: Principal Investigator, Markku Haapamaki, Associate professor, MD, PhD, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSIN-05-178M
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Pilonidal Sinus
Keywords: Sinus, Pilonidal; Pilonidal sinus; Pilonidal cysts; Pilonidal disease; midline excision; Karydakis operation; expertise based study; surgery; therapy
MeSH Terms: conditions — Pilonidal Sinus | interventions — Surgical Procedures, Operative

ARMS (2):
- Midline excision (Active Comparator): Midline excision for pilonidal sinus disease.
  Interventions: Procedure: Surgery for pilonidal disease, midline excision
- Karydakis (Active Comparator): Karydakis operation for pilonidal sinus disease.
  Interventions: Procedure: Surgery for pilonidal disease, Karydakis operation

INTERVENTIONS:
Procedure: Surgery for pilonidal disease, midline excision — A midline excision is made for the treatment of pilonidal sinus disease.
  Arms: Midline excision
Procedure: Surgery for pilonidal disease, Karydakis operation — A Karydakis operation is done for the treatment of pilonidal sinus disease.
  Arms: Karydakis

SUMMARY:
The trial compares excision in the midline at surgery for pilonidal disease versus excision lateral of the midline (Karydakis operation) at surgery for pilonidal disease by randomly allocating patients with pilonidal disease to two groups of surgeons, each group being trained for one of the two methods.

DETAILED DESCRIPTION:
Excision in the midline and primary suture is a long proven method of treating pilonidal sinus. However it's associated with high incidence of post operative infection and recurrence. On the other hand Karydakis operation (excision lateral of the midline, transposition flap and primary suture) is just a slightly more complicated procedure but has five times less recurrences reported in case series. The purpose of the present study is to compare the surgical results and costs of the two surgical methods utilized. In addition the investigators aim to compare the quality of life at defined time points after surgery. Eligible patients are randomized to two groups of surgeons, well trained in either the midline operation or the Karydakis operation (expertise based design). The design of the study allows wide inclusion criteria for participants, a cost-utility approach in the analysis, and a high external validity of the conclusions reached.

Comparison: Midline excision andd primary suture compared with the Karydakis operation (excision lateral of the midline and primary suture) for pilonidal disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Surgery is considered the best available treatment.
* The patient understands trial information and is capable of making a decision for informed consent after having received information.
* The patient wants to undergo surgery for pilonidal sinus and accepts participation in the trial.

Exclusion Criteria:

* Patient has had a pilonidal abscess during the last four weeks before the planned day of surgery
* Patient has had surgery (excision) for pilonidal sinus more than once before.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-03; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
time to complete wound healing | one year or until reoperation

SECONDARY OUTCOMES:
health-related quality of life | one year
time needed returning to normal physical activity after operation | one year or until reoperation
days spent on sick-leave | one year or until reoperation
health care costs and total costs | one year
postoperative wound infection rate | one year or until reoperation
recurrence rate | one year or until reoperation

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Odensten, MD, Principal Investigator — County Council of Norrbotten, Sweden; Markku M Haapamaki, MD, PhD, Principal Investigator — Umeå University; Peter Naredi, MD, Ph D, Study Chair — Umeå University; Michael Dahlberg, MD, PhD, Study Director — County Council of Norrbotten
Locations (2):
- Sweden (2):
  - Sunderby Regional Hospital, Luleå
  - Umeå University Hospital, Umeå

REFERENCES:
- [Background] Devereaux PJ, Bhandari M, Clarke M, Montori VM, Cook DJ, Yusuf S, Sackett DL, Cina CS, Walter SD, Haynes B, Schunemann HJ, Norman GR, Guyatt GH. Need for expertise based randomised controlled trials. BMJ. 2005 Jan 8;330(7482):88. doi: 10.1136/bmj.330.7482.88. PMID 15637373
- [Background] Petersen S, Koch R, Stelzner S, Wendlandt TP, Ludwig K. Primary closure techniques in chronic pilonidal sinus: a survey of the results of different surgical approaches. Dis Colon Rectum. 2002 Nov;45(11):1458-67. doi: 10.1007/s10350-004-6451-2. PMID 12432292
- [Background] Karydakis GE. New approach to the problem of pilonidal sinus. Lancet. 1973 Dec 22;2(7843):1414-5. doi: 10.1016/s0140-6736(73)92803-1. No abstract available. PMID 4128725
- [Background] Dalenback J, Magnusson O, Wedel N, Rimback G. Prospective follow-up after ambulatory plain midline excision of pilonidal sinus and primary suture under local anaesthesia--efficient, sufficient, and persistent. Colorectal Dis. 2004 Nov;6(6):488-93. doi: 10.1111/j.1463-1318.2004.00693.x. PMID 15521941
- [Derived] Hemmingsson O, Binnermark F, Odensten C, Rutegard M, Franklin KA, Haapamaki MM. Excision and suture in the midline versus Karydakis flap surgery for pilonidal sinus: randomized clinical trial. BJS Open. 2022 Mar 8;6(2):zrac007. doi: 10.1093/bjsopen/zrac007. PMID 35289848